CLINICAL TRIAL: NCT01914198
Title: Revisiting Parental Survey for Screening for Obstructive Sleep Apnea in Patients Undergoing Polysomnography
Status: Completed | Type: Observational
Sponsor: Vidya Raman (Other)
Responsible Party: Sponsor-Investigator, Vidya Raman, Assistant Clinical Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00338
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Sleep Apnea
Keywords: sleep study; NCH
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sleep study: Patients who are having a sleep study done at NCH to diagnose sleep apnea.
  Interventions: Other: Sleep apnea symptom survey

INTERVENTIONS:
Other: Sleep apnea symptom survey — Parents or caregivers will complete a questionnaire regarding possible sleep apnea symptoms.

SUMMARY:
The investigators are proposing a study where the investigators would give a survey to the parents of patients having a sleep study. The survey would contain questions relating to symptoms of sleep apnea and then the investigators would correlate the parent answers to the results of the sleep study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient coming for sleep study at Nationwide Children's Hospital and parent willing to fill out questionnaire.
* Children ages 3-18 years old regardless of sex or race.

Exclusion Criteria:

* Parental refusal.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are having a sleep study at NCH.
Sampling Method: Non-Probability Sample
Enrollment: 948 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

PRIMARY OUTCOMES:
Sleep apnea symptoms | 1 Day
  Parents or caregivers will be asked to complete a questionnaire regarding possible symptoms related to sleep apnea.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States